CLINICAL TRIAL: NCT05262608
Title: A Multi-center, Single-arm, Prospective Study to Investigate the Efficacy and Safety of Olaparib Monotherapy in Newly Diagnosed mCRPC Patients Who Progressed on NHA and With HRR Gene Mutation
Brief Title: The Study of Olaparib in Newly Diagnosed mCRPC Patients With HRR Gene Mutation
Acronym: PROspect
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KY-057
Record Dates: First submitted 2022-02-08; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer; Prostate Carcinoma; Metastatic Castration-resistant Prostate Cancer
Keywords: HRR; Olaparib; mCRPC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention/Treatment (Experimental): Subjects will receive a regimen of Olaparib tablets 300 mg twice daily until radiographic disease progression (assessed by the investigator according to RECIST1.1 and PCWG 3) or intolerable adverse events (assessed by the investigator according to the actual clinical situation).
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Lynparza (Olaparib tablets) 300 mg should be taken orally twice daily

SUMMARY:
This is a multi-center, single-arm, prospective study to assess the efficacy and safety of Olaparib in men with newly diagnosed metastatic castration-resistant prostate cancer (mCRPC) who carried homologous recombination repair (HRR) gene mutations and have progressed after treatment with novel endocrine agents (NHA) in the metastatic castration-sensitive prostate cancer or non-metastatic castration-resistant prostate cancer.

A total of 30 newly diagnosed mCRPC subjects with radiologically evaluable disease at baseline who have progressed on prior NHA and carry HRR gene mutations that meet the criteria will be included in the study. Eligible subjects will receive a treatment regimen of oral Olaparib tablets 300 mg twice daily until disease progression or intolerance. During the treatment and follow-up periods, all subjects will have regular visits to assess the efficacy and safety of Olaparib. Data on objective radiographic response (ORR), prostate-specific antigen response (PSA response), radiographic progression-free survival (rPFS), and time to prostate-specific antigen progression (TTPP) will be collected during the study.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, subjects should fulfil the following criteria based on local regulations:

1. Provision of informed consent prior to any study specific procedures.
2. Adult male patients (age≥18 years old).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
4. Histologically confirmed adenocarcinoma of the prostate.
5. Subjects must have previously received NHA (e.g., abiraterone acetate and/or enzalutamide) for mHSPC or nmCRPC and have disease progression to mCRPC. Disease progression was determined by the local investigator based on the diagnostic criteria for mCRPC (CRPC diagnostic criteria: testosterone maintained at castrate levels (testosterone levels less than 50 ng/dL or 1.7 nmol/L) while meeting at least one of the following criteria: A. biochemical progression: three consecutive rising PSA with an interval of at least one week between the two tests, more than 50% increase from the nadir, and PSA > 2 ng/mL; B. radiographic progression: new lesions: two or more new bone lesions on bone scan or one soft tissue lesion meeting the RECIST criteria. Symptomatic progression alone is not sufficient to diagnose CRPC. Established radiographic evidence of metastatic disease in addition to CRPC to confirm the diagnosis of mCRPC).
6. The subject had a serum testosterone level ≤ 50 ng/dL (≤ 1.75 nmol/L) before enrollment.
7. Patients who have not undergone previous surgery must be taking and voluntarily continue taking LHRH analogues (agonists or antagonists) throughout the study treatment period.
8. Subjects must have at least 1 measurable lesion at baseline (according to RECIST 1.1 criteria: At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements).
9. Subjects must have at least 1 qualifying HRR gene mutation in tumor tissue and/or plasma ct-DNA confirmed by central lab (Glorious Med, shanghai, China)

   * Archival or new biopsies are acceptable.
   * Qualifying HRR gene mutations (deleterious or suspected deleterious gene alterations) are BRCA1, BRCA2, ATM, BARD1, BRIP1, CDK12, CHEK1, CHEK2, FANCL, PALB2, RAD51B, RAD 51C, RAD51D and RAD54L mutations confirmed by the central lab.
10. Subjects must have normal organ and bone marrow function at baseline, as defined below:

    * Hemoglobin ≥ 10.0 g/dL without previous transfusion.
    * Absolute neutrophil count ≥ 1.5 × 10^9/L.
    * Platelet count ≥ 100 × 10^9/L.
    * Total bilirubin ≤ 1.5 × the upper limit of normal (ULN) specified.
    * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase/alanine aminotransferase (ALT) serum glutamic pyruvic transaminase) ≤ 2.5 × the specified ULN, unless liver metastases are present, in which case it must be ≤ 5 × ULN.
    * Estimated creatinine clearance ≥ 51 mL/min (estimated creatinine clearance = [140 - age (years)] × weight (kg)/serum creatinine (mg/dL)/72).
11. Male subject has been surgically sterilized or uses an acceptable method of contraception (defined as a barrier method with spermicide) to prevent pregnancy during the duration of the study and for 12 weeks after the dose of prednisone.
12. Subjects must have a life expectancy ≥ 16 weeks.
13. The subjects must volunteer and be capable of complying with the protocol for the duration of the study, including receiving treatment, attending scheduled visits and hospital examinations.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site) .
2. Previous enrolment in the present study.
3. Subjects participated in another clinical study with a drug or plan to participate in another interventional clinical study within 30 days prior to enrollment.
4. Prior treatment with any PARP inhibitor including Olaparib.
5. Prior chemotherapy with any DNA-damaging cytotoxic agent unless used to treat non-prostate cancer and the last dose was at least 5 years prior to enrollment in this study. For example: Patients previously treated with mitoxantrone or platinum-based chemotherapy for prostate cancer are excluded.
6. Other malignancies within the last 5 years.
7. Uncontrolled or underlying cardiac disease on resting electrocardiogram (eg, but not limited to: unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QT prolongation > 500 ms with Fridericia correction, congenital long QT syndrome).
8. The subject had received any systemic anticancer therapy (except radiotherapy) 3 weeks prior to study treatment.

   Medications used to maintain castrate status were permitted as described in Inclusion Criteria 7. Drugs such as 5-α reductase inhibitors (finasteride, dutasteride), estrogen compounds, and megestrol are considered as anticancer drugs and are prohibited at least 3 weeks before study treatment.

   Treatment of bone metastases with denosumab or bisphosphonates such as zoledronic acid is allowed.
9. Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, ritonavir, or carbidetex-boosted protease inhibitors, indinavir, saquinavir, nelfinavir, baprevir, teicoplanavir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, sulfadiazine, fluconazole, vilapamil) requires a 2-week washout period prior to initiation of Olaparib therapy.
10. Concomitant use of strong CYP3A inducers (e.g. phenobarbital, empagliflozin, phenytoin, rifampin, rifampin, rifampin, rifapentine, carbamazepine, nevirapine, and Forsythia leaf) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). If co-administered with phenobarbital, a 5-week washout period is required before the start of Olaparib therapy and a 3-week washout period is required when co-administered with other drugs.
11. Subjects with major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
12. Subjects with previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
13. Long-term toxicity (CTCAE > grade 2) due to prior cancer therapy, excluding toxicity due to alopecia or use of LHRH agonists or antagonists.
14. Subjects with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML
15. Subjects with known brain metastases (confirmation of absence of brain metastases by scan is not required).
16. Subjects with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 4 weeks.
17. Subjects who are unable to swallow oral medication and/or have a gastrointestinal disorder that would interfere with absorption of the study drug.
18. Subjects with known hypersensitivity to Olaparib or any of the excipients of this product.
19. Immunocompromised subjects, such as those with positive human immunodeficiency virus (HIV) serology.
20. Subjects with known active hepatitis (e.g. hepatitis B or C).
21. The subject has a serious, uncontrolled medical condition or non-malignant systemic disease, or an uncontrolled active infection. ( For example, but not limited to: uncontrolled arrhythmia, 12 myocardial infarction, uncontrolled seizures, extensive interstitial lung disease in both lungs, or psychiatric disease that would preclude informed consent.)-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2024-02-26 (Estimated); Study Completion 2024-04-26 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measures 1 | up to 60 months
  1. To assess the efficacy of Olaparib in newly diagnosed metastatic castration-resistant prostate cancer with mutations in homologous recombination repair genes that have progressed after prior treatment with novel endocrine agents.
  -The Overall response rate will be based on the following outcome definitions and a patient will be considered a response if any of these occur:
  (1) Objective response (ORR) according to RECIST 1.1 (soft tissue)
Primary Outcome Measures 2 | up to 60 months
  Objective response (ORR) according to PCWG-3 (bone) criteria as determined by the local investigator
Primary Outcome Measures 3 | up to 60 months
  PSA response will be reported in ng/mL (≥ 50% reduction in PSA from baseline) according to PCWG 3 criteria as determined by the local investigator

SECONDARY OUTCOMES:
Secondary Outcome Measures 1 | up to 60 months
  Investigator-assessed confirmed radiographic progression-free survival (rPFS) will be reported in weeks per RECIST 1.1 (soft tissue) and PCWG3 (bone)
Secondary Outcome Measures 2 | up to 60 months
  Investigator-assessed confirmed disease control rate (DCR) per RECIST 1.1 (soft tissue) and PCWG3 (bone)
Secondary Outcome Measures 3 | up to 60 months
  Investigator-assessed confirmed the time to PSA progression (TTPP) per PCWG3
Secondary Outcome Measures 3 | up to 60 months
  2. To assess the safety and tolerability of Olaparib in newly diagnosed metastatic castration-resistant prostate cancer with homologous recombination repair gene mutations that have progressed after prior treatment with novel endocrine agent.
  -Adverse events/Serious adverse events/AE of special interest

OTHER OUTCOMES:
Other Outcome Measures | up to 60 months
  To explore the concordance rate of tissue samples and plasma ct-DNA samples by second-generation sequencing (NGS) testing
  -Concordance rate between tissue and plasma ct-DNA testing results

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, China